CLINICAL TRIAL: NCT05906836
Title: Phase 1, Open-Label, Drug Interaction Study to Investigate the Effect of Single Dose Selpercatinib on the Pharmacokinetics of Rosuvastatin in Healthy Participants
Brief Title: A Drug Drug Interaction (DDI) Study of Selpercatinib (LY3527723) and Rosuvastatin in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: 18727; J2G-MC-JZPB (Other: Eli Lilly and Company)
Record Dates: First submitted 2023-06-08; First posted 2023-06-18 (Actual); Results first posted 2025-09-16 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-08

CONDITIONS: Healthy
Keywords: Drug Drug Interaction Trial; Selpercatinib (Retevmo®)
MeSH Terms: interventions — Rosuvastatin Calcium; selpercatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Rosuvastatin + Selpercatinib (Experimental): Participants received 20 milligram (mg) of rosuvastatin administered orally on Day 1, followed by 20 mg of rosuvastatin coadministered orally with 160 mg of selpercatinib on Day 5.
  Interventions: Drug: Rosuvastatin; Drug: Selpercatinib

INTERVENTIONS:
Drug: Rosuvastatin — Administered orally.
Drug: Selpercatinib — Administered orally.
  Other Names: LY3527723; LOXO-292; Retevmo®

SUMMARY:
The main purpose of this study is to determine the effect of selpercatinib on the levels of rosuvastatin in the blood stream in healthy participants. This study also evaluated the safety and tolerability of rosuvastatin when administered in combination with selpercatinib in healthy participants. This study will last up to approximately 26 days excluding screening period.

ELIGIBILITY:
Inclusion Criteria:

* Participants who are overtly healthy as determined by medical evaluation
* Participant must be Caucasian
* Body mass index (BMI) within the range of 19.0 to 32.0 kilograms per meter squared (kg/m²)

Exclusion Criteria:

* Have known allergies to selpercatinib-related compounds or any components of the formulation of selpercatinib, or or rosuvastatin
* • Have a significant previous or current history or presence of cardiovascular, respiratory, renal, gastrointestinal, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; of constituting a risk when taking the investigational product
* Have used or are intending to use over-the-counter or prescription medication, including dietary supplements and herbal medications, within 14 days prior to dosing

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2023-07-27 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Labcorp Clinical Research LP, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Rosuvastatin + Selpercatinib: Participants received 20 milligrams (mg) of rosuvastatin administered orally on Day 1, followed by 20 mg of rosuvastatin co-administered orally with 160 mg of selpercatinib on Day 5.
Period: Overall Study
Arm/Group | Rosuvastatin + Selpercatinib
Started | 28
Completed | 26
Not Completed | 2
Not completed — Unwilling to Make Travel Arrangements | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Population: All enrolled participants.
Groups:
- Rosuvastatin + Selpercatinib: Participants received 20 mg of rosuvastatin administered orally on Day 1, followed by 20 mg of rosuvastatin co-administered orally with 160 mg of selpercatinib on Day 5.
Arm/Group | Rosuvastatin + Selpercatinib
Number analyzed (Participants) | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.5 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10
  Not Hispanic or Latino | 18
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 27
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 28

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics (PK): Maximum Concentration (Cmax) of Rosuvastatin
Description: PK: Cmax of Rosuvastatin was reported.
Time Frame: Day 1 and Day 5: Predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, and 72 hours (h) post dose
Population: All participants who received atleast one dose of rosuvastatin and had evaluable PK data for this outcome.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per millilitre (ng/mL)
Groups:
- Rosuvastatin: Participants received 20 mg of rosuvastatin administered orally on Day 1.
- Rosuvastatin + Selpercatinib: Participants received 20 mg of rosuvastatin co-administered orally with 160 mg of selpercatinib on Day 5.
Arm/Group | Rosuvastatin | Rosuvastatin + Selpercatinib
Number analyzed (Participants) | 27 | 28
nanogram per millilitre (ng/mL) | 8.92 (59) | 15.2 (38)

2. Primary Outcome: PK: Area Under the Concentration Versus Time Curve From Time Zero to Infinity (AUC[0-∞]) of Rosuvastatin
Description: PK: AUC(0-∞) of Rosuvastatin was reported.
Time Frame: Day 1 and Day 5: Predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, and 72 h post dose
Population: All participants who received atleast one dose of rosuvastatin and had evaluable PK data for this outcome.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*hr/mL)
Arm/Group | Rosuvastatin | Rosuvastatin + Selpercatinib
Number analyzed (Participants) | 23 | 26
nanogram*hour per milliliter (ng*hr/mL) | 81.9 (70) | 151 (44)

ADVERSE EVENTS:
Time Frame: Baseline Up to Day 15
Description: All participants who received at least one dose of study drug. Based on the planned safety analysis, adverse events were collected per study treatment received.
Arm/Group | Rosuvastatin | Rosuvastatin + Selpercatinib
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/28
Other Adverse Events (participants affected / at risk) | 0/28 | 0/28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2023-05-19): https://cdn.clinicaltrials.gov/large-docs/36/NCT05906836/Prot_000.pdf
  • Statistical Analysis Plan (2023-05-24): https://cdn.clinicaltrials.gov/large-docs/36/NCT05906836/SAP_001.pdf